CLINICAL TRIAL: NCT04123860
Title: Comparative Study Between Effect of Buccal Fat Pad and Platelet Rich Fibrin After Ultrasonic Hydrodynamic Maxillary Sinus Membrane Elevation
Brief Title: Effect of Buccal Fat Pad and Platelet Rich Fibrin After Ultrasonic Hydrodynamic Maxillary Sinus Membrane Elevation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mostafa elmasry, teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: oral surgery 14
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Maxillary Sinus
Keywords: intralift; maxillery sinus lift; hydrodynamic ultrasonic; buccal pad fat; platelet rich fibrin; immediate dental implant

STUDY DESIGN:
Intervention Model Description: it is randomized clinical trail
Who Masked: Participant
Masking Description: double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- buccal fat pad (Experimental): will undergo sinus lifting using intralift technique then placement of buccal fat pad followed by immediate implant placement.
  Interventions: Other: ultrasonic hydrodynamic maxillary sinus lift buccal pad fat
- prf (Active Comparator): will undergo sinus lifting using intralift technique the prpration of PRF and immediate implant placement.
  Interventions: Other: ultrasonic hydrodynamic maxillary sinus lift platelet rich fibrin

INTERVENTIONS:
Other: ultrasonic hydrodynamic maxillary sinus lift buccal pad fat — ultrasonic hydrodynamic maxillary sinus lift and buccal fat pad as grafting material followed by immediate implant
  Other Names: intralift technique maxillary sinus lift
  Arms: buccal fat pad
Other: ultrasonic hydrodynamic maxillary sinus lift platelet rich fibrin — ultrasonic hydrodynamic maxillary sinus lift and platelet rich fibrin as grafting material followed by immediate implant
  Other Names: intralift technique maxillary sinus lift
  Arms: prf

SUMMARY:
Placing implants in the posterior maxillary area has the drawback of working with scarce, poor quality bone in a significant percentage of cases. Numerous advanced surgical techniques have been developed to overcome the difficulties associated with these limitations. Subsequent to reports on the elevation of the maxillary sinus through the lateral approach, there were reports on the use of the crestal approach, which is less aggressive but requires a minimal amount of bone. Furthermore, it is more sensitive to operator technique, as the integrity of the sinus membrane is checked indirectly. The main advantage of this new technique, Intralift, is that it does not require a minimum amount of crestal bone (indeed, the smaller the width of the crestal bone, the better this technique is performed). The possibility of damage to the sinus membrane is minimized by using ultrasound based hydrodynamic pressure to lift it, while applying a very non-aggressive crestal approach. Conclusions: We believe that this technique is an advance in the search for less traumatic and aggressive techniques, which is the hallmark of current surgery The buccal fat pad appears at 3 months in utero and continuously grows until birth (9). It protrudes at the anterior border of the masseter muscle and extends to the parotid duct, where it rests on the buccopharyngeal fascia, which covers the buccinator muscle. There is little change in the volume of buccal fat during aging, and it is approximately 10 mL

PRF is a natural fibrin-based biomaterial prepared from an anticoagulant-free blood harvest without any artificial biochemical modification that allows obtaining fibrin membranes enriched with platelets and growth factors

DETAILED DESCRIPTION:
Placing implants in the posterior maxillary area has the drawback of working with scarce, poor quality bone in a significant percentage of cases. Numerous advanced surgical techniques have been developed to overcome the difficulties associated with these limitations. Subsequent to reports on the elevation of the maxillary sinus through the lateral approach, there were reports on the use of the crestal approach, which is less aggressive but requires a minimal amount of bone. Furthermore, it is more sensitive to operator technique, as the integrity of the sinus membrane is checked indirectly. The main advantage of this new technique, Intralift, is that it does not require a minimum amount of crestal bone (indeed, the smaller the width of the crestal bone, the better this technique is performed). The possibility of damage to the sinus membrane is minimized by using ultrasound based hydrodynamic pressure to lift it, while applying a very non-aggressive crestal approach. Conclusions: We believe that this technique is an advance in the search for less traumatic and aggressive techniques, which is the hallmark of current surgery The buccal fat pad appears at 3 months in utero and continuously grows until birth (9). It protrudes at the anterior border of the masseter muscle and extends to the parotid duct, where it rests on the buccopharyngeal fascia, which covers the buccinator muscle. There is little change in the volume of buccal fat during aging, and it is approximately 10 mL

PRF is a natural fibrin-based biomaterial prepared from an anticoagulant-free blood harvest without any artificial biochemical modification that allows obtaining fibrin membranes enriched with platelets and growth factors

Sinus lifting procedures are performed routinely to provide the required height of proper and stable bone tissue around the dental implants to be inserted. The surgical technique of maxillary sinus Schneiderian membrane (MSSM) lifting with immediate/simultaneous installation of dental implants, generally results in significant bone formation. The recently reported graftless MSSM elevation procedure and the subsequent augmentation of bone have greatly changed our perspective of bone neoformation potential. The blood clot formed under the lifted MSSM appears to be of critical importance in bone neoformation potential, precluding the need for exogenous graft materials

In elevation with the rotary technique, the main intraoperative complication is perforation of Schneider's membrane, which is observed in between 10-35% of all such operations , and which usually occurs in the osteotomy drilling phase while preparing the window for access to the sinus . With the purpose of reducing the risk of perforating Schneider's membrane, vestibule osteotomy using ultrasound has been proposed, as this reduces the risk of soft tissue damage and percentage membrane perforation to 7%. Some studies in the literature are preliminary descriptions of the technique, while others present isolated cases and others in turn report case series - no significant differences being observed between the two techniques

ELIGIBILITY:
Inclusion Criteria:

* edentulous maxilla in premolar-molar areas with a residual ridge height of 5-9mm.

Exclusion Criteria:

* sinuses with septa in the operated area, polyps, sequelae of fistulas or fractures.

Cases for current study will be selected free from local pathosis. Patients will be free from any systemic disease that could affect their reparative power.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-11-10 (Estimated); Primary Completion 2020-12-10 (Estimated); Study Completion 2021-12-10 (Estimated)

PRIMARY OUTCOMES:
bone height gain | 6 month
  amount of bone gain

SECONDARY OUTCOMES:
bone density | 6 month
  change in bone density

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Sa El Hadidy, phd, Study Chair — Cairo University; Basma Ga Mousa, phd, Study Chair — Cairo University; Alaa Sh Emara, phd, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided
i will check with my study chair

REFERENCES:
- [Background] Kim MK, Han W, Kim SG. The use of the buccal fat pad flap for oral reconstruction. Maxillofac Plast Reconstr Surg. 2017 Feb 25;39(1):5. doi: 10.1186/s40902-017-0105-5. eCollection 2017 Dec. PMID 28286743
- [Background] Lo Giudice G, Iannello G, Terranova A, Lo Giudice R, Pantaleo G, Cicciu M. Transcrestal Sinus Lift Procedure Approaching Atrophic Maxillary Ridge: A 60-Month Clinical and Radiological Follow-Up Evaluation. Int J Dent. 2015;2015:261652. doi: 10.1155/2015/261652. Epub 2015 Sep 16. PMID 26451145
- [Background] Kumar KR, Genmorgan K, Abdul Rahman SM, Rajan MA, Kumar TA, Prasad VS. Role of plasma-rich fibrin in oral surgery. J Pharm Bioallied Sci. 2016 Oct;8(Suppl 1):S36-S38. doi: 10.4103/0975-7406.191963. PMID 27829743
- [Background] Velazquez-Cayon R, Romero-Ruiz MM, Torres-Lagares D, Perez-Dorao B, Wainwright M, Abalos-Labruzzi C, Gutierrez-Perez JL. Hydrodynamic ultrasonic maxillary sinus lift: review of a new technique and presentation of a clinical case. Med Oral Patol Oral Cir Bucal. 2012 Mar 1;17(2):e271-5. doi: 10.4317/medoral.17430. PMID 22143696
- [Background] Penarrocha-Diago M, Penarrocha-Diago M, Sanchez-Recio C, Penarrocha-Oltra D, Romero-Millan J. Osteotomy in direct sinus lift. A comparative study of the rotary technique and ultrasound. Med Oral Patol Oral Cir Bucal. 2012 May 1;17(3):e457-61. doi: 10.4317/medoral.17599. PMID 22143735